CLINICAL TRIAL: NCT04151472
Title: A Randomized, Double-blinded, Placebo-controlled Trial of Idebenone in the Prevention of Episodic Migraine
Brief Title: Idebenone for the Preventive Treatment of Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Kaiming Liu, Deputy chief physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-675
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Migraine Disorders; Headache Disorders
Keywords: Migraine Prophylaxis; Mitochondrial Dysfunction; Idebenone; Individualized Treatment
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Mitochondrial Diseases | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 90mg Idebenone (Experimental): Placebo by mouth, three times a day for 1 months； Idebenone 30mg table by mouth, three times a day for next 3 months
  Interventions: Drug: Placebo; Drug: 90mg Idebenone
- 270mg Idebenone (Experimental): Placebo by mouth, three times a day for 1 months； Idebenone 90mg table by mouth, three times a day for next 3 months
  Interventions: Drug: Placebo; Drug: 270mg Idebenone
- Placebo (Placebo Comparator): Placebo by mouth, three times a day for 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo oral tablet, three times a day
Drug: 90mg Idebenone — Idebenone 30 MG Oral Tablet, three times a day
  Other Names: Shenwei
  Arms: 90mg Idebenone
Drug: 270mg Idebenone — Idebenone 90 MG Oral Tablet, three times a day
  Other Names: Shenwei
  Arms: 270mg Idebenone

SUMMARY:
Idebenone improves energy metabolism similarly to Coenzyme Q10, which is effective in migraine prophylaxis. The investigators compare idebenone (90 mg/day, 270 mg/day) and placebo in 180 migraine patients in a double-blind, randomized, placebo-controlled, multicenter trial to study whether Idebenone is superior to placebo in the prevention of episodic migraine with or without aura.

DETAILED DESCRIPTION:
One-hundred-and-eighty subjects will be recruited for a placebo-controlled, double-blinded study of idebenone (90 mg/day, 270 mg/day) versus placebo. One-hundred-and-eighty subjects will be recruited based on past research and an expected 20% dropout rate. A dose of 90mg or 270 mg is based on large number of reports at study initiation in Leber's hereditary optic neuropathy that demonstrated the safety of 900mg/day. Subjects are 18 to 65 years old, inclusive, who meet the International Classification of Headache Disorder- III (ICHD-III) for episodic migraine with or without aura, no over consumption of acute anti-migraine medication, no other prophylactic medication (washout 3 months), no serious organic or psychiatric disease, who are recommended to start prophylactic therapy (two to eight attacks per month). Written informed consent is obtained. The process of patients through the trial phases follows the CONSORT flow chart.

Idebenone and placebo were provided by Qilu Pharmaceutical Company Limited, China. Placebo consisted of the same ingredients as verum-instead idebenone, they classify as fit for human consumption in the China and without any known effect on migraine.

The design of this double-blind, randomized, placebo-controlled trial followed the IHS Committee on Clinical Trials in Migraine guidelines, 8 current EU guidelines on Good Clinical Practice, and the Declaration of Helsinki. It was approved by Neurology Department, the Second Affiliated Hospital, School of Medicine, Zhejiang University. This study is supported by the following funding sources: the Zhejiang Provincial Natural Science Foundation of China (Grant No. LY19H090025, Grant No. LQ15H090003), the National Natural Science Foundation of China (Grant No. 81101157). The study is also supported by Qilu Pharmaceutical Company Limited, China (http://www.qilu-pharma.com); the use of idebenone in migraine, is patent pending in the China. Dr. Kaiming Liu do not receive honoraria from the sponsor of the study.

Exclusion criteria includes subjects who previously failed idebenone therapy for migraine prophylaxis, those who previously discontinued idebenone due to adverse events, those who are taking idebenone or had taken idebenone within 14 days prior to enrollment, and subjects with continuous headaches. Subjects will be equally randomized to be treated with 90 mg/day idebenone, 270 mg/day idebenone, or placebo for 3 months.

At the first visit, patients will receive placebo for a 1-month base-line. At the second visit, they will be randomized to be treated with 90 mg/day idebenone, 270 mg/day idebenone, or placebo for next 3 months if they have presented at least one migraine attack.

The primary objective is to assess whether at least 1 dose of Idebenone is superior to placebo in overall mean change from baseline of 4-week migraine headache days (MHD) during double-blind treatment. Key secondary outcome variables will be change of migraine attack frequency, migraine moderate/severe headache days, the proportion of subjects with at least 50%, at least 75%, and 100% reduction in migraine days, mean severity of migraine, acute treatment utilization, quality of life related to episodic migraine as measured by the The Role Function Physical subscale in The Migraine-Specific Quality of Life questionnaire (MSQ v2.1), migraine-related disability as measured by The Headache Impact Test (HIT-6), Patient Global Impression of Severity (PGI-S) scores, and Migraine Disability Assessment (MIDAS) scores from baseline of 4-week to the entire double-blind treatment phase.

Responders for attack frequency (50% reduction) will be calculated and the number-needed-to-treat (NNT) determined. Patients will be interviewed about adverse events at each visit. Statistical analysis will be done on an intention-to-treat population applying the last visit carried forward method. Mann-Whitney U test will be used for differences between groups, 2 test for 22 contingency tables of responder rate, general linear mixed model for evolution over time. Significance level is p<0.05, after accounting for multiple comparisons. SPSS will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of episodic migraine.
2. Patients (18-65 years) were eligible if they met International Headache Society (IHS) criteria for episodic migraine with/ without aura with a migraine history 1 year
3. Two to eight attacks per month, 5 days/month of interval headaches.
4. No over consumption of acute anti-migraine medication.
5. No other prophylactic medication (washout 3 months).
6. No serious organic or psychiatric disease.
7. Only women with contraceptive protection.

Exclusion Criteria:

1. Clinical diagnosis of chronic migraine.
2. Subjects previously discontinued idebenone due to adverse events.
3. Subjects are taking idebenone or had taken idebenone within 14 days prior to enrollment.
4. Subjects with continuous headaches.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of migraine attack frequency | month 0, month 1, month 2, month 3, month 4
  The change of migraine attack frequency in month 4 compared with baseline. Headache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary. Degree of pain and results of treatment are scored by visual analogue scale(VAS).

SECONDARY OUTCOMES:
The change of days with headache | month 0, month 1, month 2, month 3, month 4
  The change of days with headache per month compared with baseline. Headache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary.
Mean severity of migraine | month 0, month 1, month 2, month 3, month 4
  Mean severity of migraine per month compared with baselineHeadache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary. Degree of pain is scored by VAS.
The change of days with nausea/vomiting | month 0, month 1, month 2, month 3, month 4
  The change of days with nausea/vomiting per month compared with baselineHeadache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary.
Mean duration of migraine | month 0, month 1, month 2, month 3, month 4
  Mean duration of migraine per month compared with baselineHeadache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary.
50% Responder rate for attack frequency | month 0, month 1, month 2, month 3, month 4
  50% Responder rate for attack frequency compared with baselineHeadache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary.
Mean no. tablets per day | month 0, month 1, month 2, month 3, month 4
  Mean no. tablets per day compared with baselineHeadache data (e.g., occurrence, duration, and pain severity; occurrence of photophobia, phonophobia, nausea, or vomiting; and any use of migraine medication) were captured daily through a daily headache-diary.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiming Liu, MD & PHD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Kaiming Liu, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Some subjects do not hope that their IPD are used by other researchers.

REFERENCES:
- [Background] Dalla Volta G, Carli D, Zavarise P, Ngonga G, Vollaro S. P026. Pilot study on the use of coenzyme Q10 in a group of patients with episodic migraine without aura. J Headache Pain. 2015 Dec;16(Suppl 1):A186. doi: 10.1186/1129-2377-16-S1-A186. No abstract available. PMID 28132202
- [Background] Dahri M, Tarighat-Esfanjani A, Asghari-Jafarabadi M, Hashemilar M. Oral coenzyme Q10 supplementation in patients with migraine: Effects on clinical features and inflammatory markers. Nutr Neurosci. 2019 Sep;22(9):607-615. doi: 10.1080/1028415X.2017.1421039. Epub 2018 Jan 3. PMID 29298622
- [Background] Gaul C, Diener HC, Danesch U; Migravent(R) Study Group. Improvement of migraine symptoms with a proprietary supplement containing riboflavin, magnesium and Q10: a randomized, placebo-controlled, double-blind, multicenter trial. J Headache Pain. 2015;16:516. doi: 10.1186/s10194-015-0516-6. Epub 2015 Apr 3. PMID 25916335
- [Background] Yorns WR Jr, Hardison HH. Mitochondrial dysfunction in migraine. Semin Pediatr Neurol. 2013 Sep;20(3):188-93. doi: 10.1016/j.spen.2013.09.002. PMID 24331360
- [Background] Markley HG. CoEnzyme Q10 and riboflavin: the mitochondrial connection. Headache. 2012 Oct;52 Suppl 2:81-7. doi: 10.1111/j.1526-4610.2012.02233.x. PMID 23030537
- [Background] Slater SK, Nelson TD, Kabbouche MA, LeCates SL, Horn P, Segers A, Manning P, Powers SW, Hershey AD. A randomized, double-blinded, placebo-controlled, crossover, add-on study of CoEnzyme Q10 in the prevention of pediatric and adolescent migraine. Cephalalgia. 2011 Jun;31(8):897-905. doi: 10.1177/0333102411406755. Epub 2011 May 17. PMID 21586650
- [Background] Brenner SR. Mitochondrial DNA haplogroups influence the therapeutic response to riboflavin in migraineurs. Neurology. 2010 Jan 12;74(2):182-3; author reply 183. doi: 10.1212/WNL.0b013e3181c77678. No abstract available. PMID 20065258
- [Background] Rozen TD, Oshinsky ML, Gebeline CA, Bradley KC, Young WB, Shechter AL, Silberstein SD. Open label trial of coenzyme Q10 as a migraine preventive. Cephalalgia. 2002 Mar;22(2):137-41. doi: 10.1046/j.1468-2982.2002.00335.x. PMID 11972582
- [Background] Borkum JM. Migraine Triggers and Oxidative Stress: A Narrative Review and Synthesis. Headache. 2016 Jan;56(1):12-35. doi: 10.1111/head.12725. Epub 2015 Dec 7. PMID 26639834
- [Background] Koreshkina MI. [The use of noben (idebenone) in the complex treatment of episodic and chronic migraine]. Zh Nevrol Psikhiatr Im S S Korsakova. 2010;110(6):98-101. No abstract available. Russian. PMID 20726168
- [Background] Klopstock T, Yu-Wai-Man P, Dimitriadis K, Rouleau J, Heck S, Bailie M, Atawan A, Chattopadhyay S, Schubert M, Garip A, Kernt M, Petraki D, Rummey C, Leinonen M, Metz G, Griffiths PG, Meier T, Chinnery PF. A randomized placebo-controlled trial of idebenone in Leber's hereditary optic neuropathy. Brain. 2011 Sep;134(Pt 9):2677-86. doi: 10.1093/brain/awr170. Epub 2011 Jul 25. PMID 21788663